CLINICAL TRIAL: NCT02425423
Title: Study on the Tolerance and Efficacy of a New Anti Regurgitation Formula
Acronym: SONAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-01-SONAR
Record Dates: First submitted 2015-04-20; First posted 2015-04-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- New thickened infant formula (Experimental)
  Interventions: Dietary Supplement: New thickened formula

INTERVENTIONS:
Dietary Supplement: New thickened formula

SUMMARY:
The aim of this study is to evaluate the efficacy of a new thickened formula on regurgitation.

ELIGIBILITY:
Inclusion Criteria:

Infants :

* Aged ≤ 5 months old
* fully formula fed
* with at least 5 episodes of regurgitation per day

Exclusion Criteria:

* Breast fed infants
* Infants presenting symptoms of a complicated gastroesophageal reflux
* Infants presenting intestinal disorders

Max Age: 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of episodes of regurgitation per day | 14 days

SECONDARY OUTCOMES:
Regurgitation score | 14 days
Regurgitation score | 3 months
Digestive tolerance (stools' number and consistency) | 14 days
  Digestive tolerance of the formula assessed through stools' number and consistency
Digestive tolerance (stools' number and consistency) | 3 months
  Digestive tolerance of the formula assessed through stools' number and consistency
Growth parameters (Weight, height and head circumference) | 3 months
  Weight, height and head circumference

CONTACTS AND LOCATIONS:
Overall Officials: Yvan Vandenplas, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (3):
- Belgium (2):
  - Pediatricians, Belgium
  - Universitair Ziekenhuis, Brussels
- Pediatricians, France, France